CLINICAL TRIAL: NCT00918307
Title: Comparison of the Efficacy and Safety of Varenicline Versus Placebo for Smoking Cessation Among HIV-infected Patients. A Randomized Double Blind Controlled Trial
Brief Title: Efficacy and Safety of Varenicline Among HIV-infected Patients
Acronym: Inter-ACTIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-007948-34; ANRS 144
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infections; Tobacco Dependence
Keywords: Tobacco Dependence; HIV infection; varenicline
MeSH Terms: conditions — HIV Infections; Tobacco Use Disorder | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Experimental): Varenicline titrated to 2 x 0.5 mg twice daily for 12 weeks
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): placebo titrated to 2 pills twice daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Day 1 to day 3 : 0.5 mg daily ; Day 4 to day 7 : 0.5 mg twice daily ; Day 8 to week 12 : 2 x 0.5 mg twice daily
  Other Names: Champix
  Arms: Varenicline
Drug: Placebo — Day 1 to day 3 : 1 pill daily ; Day 4 to day 7 : 2 pills daily ; Day 8 to week 12 : 2 pills twice daily
  Arms: Placebo

SUMMARY:
Cigarette smoking is a major cause of illness among HIV-infected patients (non-AIDS defining malignancies (especially lung cancer), non-AIDS bacterial infections and cardio-vascular diseases). Approximately 50% of HIV-infected patients are regular tobacco smokers. Tobacco smoking cessation has well known benefits on mortality and morbidity in the general population where tobacco cessation assistance programs are increasingly implemented. However, smoking cessation interventions have never been evaluated among HIV-infected patients. This trial aims at evaluating the efficacy and safety of varenicline for smoking cessation compared with placebo.

DETAILED DESCRIPTION:
Cigarette smoking is a major cause of illness among HIV-infected patients (non-AIDS defining malignancies (especially lung cancer), non-AIDS bacterial infections and cardio-vascular diseases). Approximately 50% of HIV-infected patients are regular tobacco smokers. Tobacco smoking cessation has well known benefits on mortality and morbidity in the general population where tobacco cessation assistance programs are increasingly implemented. However, smoking cessation interventions have never been evaluated among HIV-infected patients. This trial aims at evaluating the efficacy and safety of varenicline for smoking cessation compared with placebo. A pharmacokinetic study will be conducted to evaluate the effect of smoking cessation on the plasma concentration of antiretroviral treatment.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients
* adults
* regular smokers (at least 10 cigarettes a day during the last year)
* motivated to stop smoking
* followed in one of the participating clinical ward,
* signed written inform consent

Exclusion Criteria:

* current co-dependency to another psychoactive substance
* ongoing depressive episode
* history of suicidal attempt
* ongoing treatment by interferon
* treatment by efavirenz for less than three months or not tolerated
* previous use of varenicline
* ongoing treatment by bupropion-SR or nicotinic substitute
* ongoing pregnancy
* ongoing breastfeeding
* hypersensitivity to varenicline or to one of its excipients
* drivers, air traffic controller

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2009-10; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Continuous abstinence from smoking from week 9 to week 48 without the use of any other smoking cessation treatments other than trials' treatment | from week 9 to week 48

SECONDARY OUTCOMES:
Continuous abstinence from smoking from week 9 to week 12 without the use of any other smoking cessation treatments other than trials' treatment | from week 9 to week 12
Change in Lung capacity (FEV1 and FVC) between inclusion and week 48 | week 48
Frequency of depressive episodes. Diagnosed by a psychiatrist | continuously
Change in cardiovascular risk score (Framingham and PROCAM scores) between inclusion and week 48. | week 48
Quality of life evaluation (SF-12) | inclusion, W12, W24, W48

CONTACTS AND LOCATIONS:
Overall Officials: Patrick MERCIE, MD, Principal Investigator — CHU de Bordeaux, F-33000; Geneviève CHENE, MD, PHD, Study Chair — INSERM U897
Locations (1):
- CHU de Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Mdege ND, Shah S, Dogar O, Pool ER, Weatherburn P, Siddiqi K, Zyambo C, Livingstone-Banks J. Interventions for tobacco use cessation in people living with HIV. Cochrane Database Syst Rev. 2024 Aug 5;8(8):CD011120. doi: 10.1002/14651858.CD011120.pub3. PMID 39101506
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Mercie P, Arsandaux J, Katlama C, Ferret S, Beuscart A, Spadone C, Duvivier C, Reynes J, Wirth N, Moinot L, Benard A, Zucman D, Duval X, Molina JM, Spire B, Fagard C, Chene G; ANRS 144 Inter-ACTIV study group. Efficacy and safety of varenicline for smoking cessation in people living with HIV in France (ANRS 144 Inter-ACTIV): a randomised controlled phase 3 clinical trial. Lancet HIV. 2018 Mar;5(3):e126-e135. doi: 10.1016/S2352-3018(18)30002-X. Epub 2018 Jan 9. PMID 29329763
- See also: Related Info — http://www.anrs.fr